CLINICAL TRIAL: NCT00155025
Title: Family History in Prostate Cancer Patients in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700594
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2004-04

CONDITIONS: Prostate Cancer
Keywords: Prostatic neoplasms; Family history
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
To investigate the prevalence of family history in prostate cancer patients in Taiwan and evaluate the association of variation of diseases and family history

DETAILED DESCRIPTION:
We retrospectively reviewed the medical charts of prostate cancer patients at NTUH from 1978 to 2002. The initial presentations, systemic diseases, smoking habits, clinical stages, Gleason scores, pathological stages, treatments, and outcome were recorded. Post-hoc questionnaires were completed with OPD visits, admission visits, telephone interviews and mails. The questionnaires included the family histories of prostate cancer, colon cancer, breast cancer, hepatoma and so on. If patients is passed away, the first degree relatives will fill the vacant position. The prevalence of family histories of prostate cancers in these patients was determined. The associations of family histories and clinical presentations were analyzed. Besides, the characteristics of patients with and without responses were discussed.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients who were recorded at National Taiwan University Hospital from 1977 to 2002.

Exclusion Criteria:

* Patients or their family who refused our contact or were unable to be contacted

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan